CLINICAL TRIAL: NCT00000463
Title: Post Coronary Artery Bypass Graft (CABG) Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 52
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia | interventions — Lovastatin; Cholestyramine Resin; Warfarin

INTERVENTIONS:
Drug: lovastatin
Drug: cholestyramine
Drug: warfarin

SUMMARY:
To determine the relative effectiveness of moderate versus more aggressive lipid lowering, and of low dose anticoagulation versus placebo, in delaying saphenous vein coronary bypass graft atherosclerosis and preventing occlusion of saphenous grafts of patients with saphenous vein coronary bypass grafts placed 1 to 11 years previously.

DETAILED DESCRIPTION:
BACKGROUND:

A large number of studies have reported that following CABG, the vessels proximal to the grafts demonstrate accelerated atherosclerosis and the grafts themselves may show progressive obstruction due to thrombosis, fibrosis, and graft atheroma. Pathological and clinical studies have documented that graft obstruction during the perioperative period and the first year is usually due to technical problems at surgery or thrombosis and occurs in about 15 to 20 percent of saphenous vein grafts. Antiplatelet drugs such as aspirin have been shown to reduce these early graft occlusions by about 50 percent. In addition to thrombosis, during the first year, most saphenous vein grafts undergo diffuse fibrosis and some distortion. However, the significance of these changes is not known.

After the first year, lipid deposition and changes histologically similar to atherosclerosis have been documented both in experimental studies and in human saphenous vein grafts patent at one year completely occlude and an additional 30 percent narrow over a period of ten years. These angiographic changes in the saphenous vein grafts correlate with high LDL-cholesterol, low HDL-cholesterol and high apolipoprotein B levels. In experimental animals, cholesterol deposition in the grafts has been substantially increased or decreased by increasing or decreasing the saturated fats and cholesterol in the animal's diets. In contrast to changes in the saphenous vein grafts, internal mammary artery grafts have shown substantially lower rates of obstruction. The native vessels (both ungrafted vessels and grafted vessels at distal or proximal sites), however, show evidence of progressive atherosclerosis. The long-term follow-up of grafts also demonstrates thrombotic material and even occlusive thrombus as part of acute events.

Progression of atherosclerotic lesions in grafts and native vessels lead to recurrent angina, unaltered long-term survival and reduced efficacy of repeat CABG surgery. Johnson in an 11 year follow-up of 3,105 post-CABG patients, reported that about 15 percent of patients with preoperative angina have recurrent angina at 1 year; with a further 6 percent developing angina every subsequent year. In this study, patients with recurrent angina had twice the mortality compared to those who were angina-free. Long-term follow-up of the VA Cooperative Trial of CABG shows that the survival of the surgical group appears to be initially superior compared to the medical group but this benefit is diminished by about ten years. This may relate to graft obstruction and progression of native coronary atherosclerosis. Re-operation in these patients carries a higher operative mortality risk and the results are less impressive. It had been estimated that approximately 5 percent of all CABG surgery in 1984 were re-operations and that this percentage would double over the next decade. Therefore, measures to prevent graft occlusion and progression of atherosclerosis in native vessels, if successful, could have substantial clinical and economic importance by reducing mortality, morbidity and the numbers of patients undergoing re-operations.

Apart from trials of aspirin and dipyridamole in post-CABG patients that demonstrated a significant reduction in graft closure within the first year after surgery, there were no large systematic studies of interventions in these patients. Graft occlusion has been shown to correlate with high LDL-cholesterol and low HDL-cholesterol, and the severity of atherosclerosis has been additionally shown to be related to cigarette smoking and increased levels of coagulation factor. Therefore, lowering the LDL cholesterol (by diet and drugs), and anti-thrombotic therapy with warfarin were logical choices for intervention.

Several studies suggested that CABG surgery relieved angina and improved overall quality of life. However, in the available studies, CABG did not consistently appear to be associated with an improvement in employment status, physical recreational activity, or life style. The reasons for these results were not entirely clear and there was a need to identify the biobehavioral and psychosocial factors that predicted successful adjustment after CABG.

The initiative was proposed by Institute staff and approved by the September 1985 National Heart, Lung, and Blood Advisory Council. The Request for Proposals was released in September 1985 and awards made in April 1987.

DESIGN NARRATIVE:

Multicenter, double-blind, randomized, controlled trial. All prospective participants received active warfarin treatment for a month prior to randomization. Only participants demonstrating a minimal reaction to warfarin and consuming over 90 percent of the prescribed medication were randomized. Dietary modification to lower serum cholesterol, an exercise program, and a smoking cessation program were implemented. Patients were randomly assigned in a 2 X 2 factorial design in four treatment groups: aggressive LDL-C lowering with lovastatin 40 to 80 mg/d and, as necessary cholestyramine 8 mg/d to achieve and LDL-C of 60 to 85 mg/dl; moderate LDL-C lowering with lovastatin 2.5 to 5 mg/d, with cholestyramin as needed, to achieve a LDL-C of 130 to 140 mg/dl; warfarin 1 to 4 mg/d to achieve an INR of 1.8 to 2.0; and warfarin-placebo. All participants were followed for five years, at the end of which selective coronary and graft angiography was performed. The primary angiography endpoint was the proportion of major SVG per patient that showed substantial reduction (0.06 mm or greater) in lumen diameter. Biobehavioral studies were conducted in 750 participants.

Planning for the study began in April 1987 and a final protocol was developed by August 1988. Patient recruitment has been completed. Follow-up ended on September 1, 1995 and data analysis continues through December 1998 under contract N01-HC-75076. .

The Post CABG Biobehavioral Study examined a cohort of 759 coronary artery bypass patients (269 women and 490 men) who were enrolled at five clinical centers. Sociodemographic and medical data were obtained by interview and from medical charts. Health-related quality of life and psychosocial data were ascertained preoperatively by interview and questionnaire for those patients whose condition allowed preoperative assessment and was compared among patients from hospitals enrolling both male and female patients.

ELIGIBILITY:
Men and women between 1 and 11 years post-CABG. Patients had two completely independent saphenous vein grafts that were patent. Patients had an LDL-cholesterol between 130 and 175 with plasma triglycerides below 300 mg/dl.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1987-04; Study Completion 1998-12

CONTACTS AND LOCATIONS:
Overall Officials: Genell Knatterud — Maryland Medical Research Institute

REFERENCES:
- [Background] Healy B, Campeau L, Gray R, Herd JA, Hoogwerf B, Hunninghake D, Knatterud G, Stewart W, White C. Conflict-of-interest guidelines for a multicenter clinical trial of treatment after coronary-artery bypass-graft surgery. N Engl J Med. 1989 Apr 6;320(14):949-51. doi: 10.1056/NEJM198904063201432. No abstract available. PMID 2784541
- [Background] Fox NL, LoPresti F, Hoogwerf B, Knatterud G, Linquist R, Czajkowski S. Self-administered quality of life forms: experience from the Post Coronary Artery Bypass Graft Studies. Controlled Clin Trials 1993;14:402.
- [Background] Shenberger DM, Helgren RJ, Peters JR, Quiter E, Johnston EA, Hunninghake DB. Intense dietary counseling lowers LDL cholesterol in the recruitment phase of a clinical trial of men who had coronary artery bypass grafts. J Am Diet Assoc. 1992 Apr;92(4):441-5. PMID 1556345
- [Background] Campeau L, Knatterud GL, White C, Domanski M, Geller N, Robernsberg Y and the Post CABG Studies Principal Investigators. The NHLBI Post Coronary Artery Bypass Graft Clinical Trial (Post CABG): Angiographic outcomes. Proceedings of the colloquium "Progression and Regression of Coronary Atherosclerosis: Observations from Lipid Intervention Studies," In Press
- [Background] Post Coronary Artery Bypass Graft Trial Investigators. The effect of aggressive lowering of low-density lipoprotein cholesterol levels and low-dose anticoagulation on obstructive changes in saphenous-vein coronary-artery bypass grafts. N Engl J Med. 1997 Jan 16;336(3):153-62. doi: 10.1056/NEJM199701163360301. PMID 8992351
- [Background] Fuster V, Vorchheimer DA. Prevention of atherosclerosis in coronary-artery bypass grafts. N Engl J Med. 1997 Jan 16;336(3):212-3. doi: 10.1056/NEJM199701163360309. No abstract available. PMID 8988902
- [Background] Czajkowski SM, Terrin M, Lindquist R, Hoogwerf B, Dupuis G, Shumaker SA, Gray JR, Herd JA, Treat-Jacobson D, Zyzanski S, Knatterud GL. Comparison of preoperative characteristics of men and women undergoing coronary artery bypass grafting (the Post Coronary Artery Bypass Graft [CABG] Biobehavioral Study). Am J Cardiol. 1997 Apr 15;79(8):1017-24. doi: 10.1016/s0002-9149(97)00040-4. PMID 9114757
- [Background] Canner PL, Thompson B, Knatterud GL, Geller N, Campeau L, Zucker D. An application of the Zucker-Wittes modified ratio estimate statistic in the Post Coronary Artery Bypass Graft (CABG) clinical trial. Control Clin Trials. 1997 Aug;18(4):318-27. doi: 10.1016/s0197-2456(96)00232-2. PMID 9257071
- [Background] Hoogwerf BJ, Waness A, Cressman M, Canner J, Campeau L, Domanski M, Geller N, Herd A, Hickey A, Hunninghake DB, Knatterud GL, White C. Effects of aggressive cholesterol lowering and low-dose anticoagulation on clinical and angiographic outcomes in patients with diabetes: the Post Coronary Artery Bypass Graft Trial. Diabetes. 1999 Jun;48(6):1289-94. doi: 10.2337/diabetes.48.6.1289. PMID 10342818
- [Background] Gobel FL, Stewart WJ, Campeau L, Hickey A, Herd JA, Forman S, White CW, Rosenberg Y. Safety of coronary arteriography in clinically stable patients following coronary bypass surgery. Post CABG Clinical Trial Investigators. Cathet Cardiovasc Diagn. 1998 Dec;45(4):376-81. doi: 10.1002/(sici)1097-0304(199812)45:43.0.co;2-x. PMID 9863740
- [Background] Hunninghake DB. Is aggressive cholesterol control justified? Review of the post-coronary artery bypass graft trial. Am J Cardiol. 1998 Nov 26;82(10B):45T-48T. doi: 10.1016/s0002-9149(98)00725-5. PMID 9860374
- [Background] Knatterud GL, Rosenberg Y, Campeau L, Geller NL, Hunninghake DB, Forman SA, Forrester JS, Gobel FL, Herd JA, Hickey A, Hoogwerf BJ, Terrin ML, White C. Long-term effects on clinical outcomes of aggressive lowering of low-density lipoprotein cholesterol levels and low-dose anticoagulation in the post coronary artery bypass graft trial. Post CABG Investigators. Circulation. 2000 Jul 11;102(2):157-65. doi: 10.1161/01.cir.102.2.157. PMID 10889125
- [Background] Domanski MJ, Borkowf CB, Campeau L, Knatterud GL, White C, Hoogwerf B, Rosenberg Y, Geller NL. Prognostic factors for atherosclerosis progression in saphenous vein grafts: the postcoronary artery bypass graft (Post-CABG) trial. Post-CABG Trial Investigators. J Am Coll Cardiol. 2000 Nov 15;36(6):1877-83. doi: 10.1016/s0735-1097(00)00973-6. PMID 11092659
- [Background] Campeau L, Hunninghake DB, Knatterud GL, White CW, Domanski M, Forman SA, Forrester JS, Geller NL, Gobel FL, Herd JA, Hoogwerf BJ, Rosenberg Y. Aggressive cholesterol lowering delays saphenous vein graft atherosclerosis in women, the elderly, and patients with associated risk factors. NHLBI post coronary artery bypass graft clinical trial. Post CABG Trial Investigators. Circulation. 1999 Jun 29;99(25):3241-7. doi: 10.1161/01.cir.99.25.3241. PMID 10385497
- [Background] Alaupovic P, Fesmire JD, Hunnighake D, Domanski M, Forman S, Knatterud GL, Forrester J, Herd JA, Hoogwerf B, Campeau L, Gobel FL. The effect of aggressive and moderate lowering of LDL-cholesterol and low dose anticoagulation on plasma lipids, apolipoproteins and lipoprotein families in post coronary artery bypass graft trial. Atherosclerosis. 1999 Oct;146(2):369-79. doi: 10.1016/s0021-9150(99)00151-3. PMID 10532693
- [Background] White CW, Campeau L, Canner P, Domanski M, Forrester JS, Gobel FL, Herd JA, Hoogwerf BJ, Hunninghake DB, Knatterud GL, LoPresti F; Post CABG Investigators. Lessons from the post coronary artery bypass graft study in evaluating and controlling technical variability in angiographic trials. Post CABG Investigators. Am J Cardiol. 2001 Jan 1;87(1):40-3. doi: 10.1016/s0002-9149(00)01269-8. PMID 11137831
- [Background] White CW, Gobel FL, Campeau L, Knatterud GL, Forman SA, Forrester JS, Geller NL, Herd JA, Hickey A, Hoogwerf BJ, Hunninghake DB, Rosenberg Y, Terrin ML; Post Coronary Artery Bypass Graft Trial Investigators. Effect of an aggressive lipid-lowering strategy on progression of atherosclerosis in the left main coronary artery from patients in the post coronary artery bypass graft trial. Circulation. 2001 Nov 27;104(22):2660-5. doi: 10.1161/hc4701.099730. PMID 11723015
- [Background] Herd JA, Hoogwerf BJ, Barton F, Terrin ML, Czajkowski SM, Lindquist R, Dupuis G. Heart rate and blood pressure responses to mental stress and clinical cardiovascular events in men and women after coronary artery bypass grafting: the Post Coronary Artery Bypass Graft (Post-CABG) biobehavioral study. Am Heart J. 2003 Aug;146(2):273-9. doi: 10.1016/S0002-8703(03)00182-0. PMID 12891195
- [Background] Lindquist R, Dupuis G, Terrin ML, Hoogwerf B, Czajkowski S, Herd JA, Barton FB, Tracy MF, Hunninghake DB, Treat-Jacobson D, Shumaker S, Zyzanski S, Goldenberg I, Knatterud GL; POST CABG Biobehavioral Study Investigators. Comparison of health-related quality-of-life outcomes of men and women after coronary artery bypass surgery through 1 year: findings from the POST CABG Biobehavioral Study. Am Heart J. 2003 Dec;146(6):1038-44. doi: 10.1016/S0002-8703(03)00451-4. PMID 14660996
- [Background] Campeau L, Knatterud G, Hunninghake B, Domanski M. Optimizing cholesterol lowering therapy: contribution of the Post Coronary Artery Bypass Graft Trial. Eur Heart J. 1997 Nov;18(11):1683-5. doi: 10.1093/oxfordjournals.eurheartj.a015155. No abstract available. PMID 9402435
- [Background] Fox NL, Hoogwerf BJ, Czajkowski S, Lindquist R, Dupuis G, Herd JA, Campeau L, Hickey A, Barton FB, Terrin ML; POST CABG Study Investigators. Quality of life after coronary artery bypass graft: results from the POST CABG Trial. Chest. 2004 Aug;126(2):487-95. doi: 10.1378/chest.126.2.487. PMID 15302735
- Available data/document: Individual Participant Data Set: CABG — http://biolincc.nhlbi.nih.gov/studies/cabg/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.